CLINICAL TRIAL: NCT06586619
Title: A Remotely Delivered Tai Chi/Qigong Intervention for Older People Living With HIV: A Randomized Clinical Trial
Brief Title: A Remotely Delivered Tai Chi/Qigong Intervention for Older People Living With HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Arizona State University (Other); University of Miami (Other); New College of Florida (Unknown)
Responsible Party: Principal Investigator, Gladys Ibanez, PhD, Associate Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 800019107; 1R01AT012590-01A1 (NIH)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Depressive Symptoms; Hiv
Keywords: Depression; HIV; older; tai chi; mindfulness; intervention
MeSH Terms: conditions — Depression; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai chi/qigong group (Experimental): This is a behavioral intervention that consist of tai chi/qigong group classes via Zoom twice a week for 12 weeks.
  Interventions: Behavioral: Tai chi/qigong intervention group
- Health education group (Active Comparator): This is a general health education control group class that will also be delivered via Zoom and will be twice a week for 12 weeks.
  Interventions: Behavioral: Health Education group

INTERVENTIONS:
Behavioral: Tai chi/qigong intervention group — The intervention is a tai chi/qigong intervention for older people living with HIV. This behavioral group-based intervention will be delivered through Zoom twice a week for 12 weeks. Each class lasts 45-60 minutes. Tai chi/qigong is a slow low impact meditative movement.
  Arms: Tai chi/qigong group
Behavioral: Health Education group — Participants will be assigned to a health and wellness education group for older people living with HIV. This group will be delivered through Zoom twice a week for 12 weeks, and each class will last 45-60 minutes. Each group will learn about and discuss a health and wellness topic.
  Arms: Health education group

SUMMARY:
The goal of this randomized clinical trial is to learn if tai chi/qigong decreases depressive symptoms among older people living with HIV compared to a health education class. The main questions it aims to answer are:

Does tai chi/qigong reduce depressive symptoms among older people living with HIV more than a health education class? What are the behavioral, psychological, and biological mechanisms in which tai chi/qigong affects depressive symptoms? Does tai chi/qigong affect depressive symptoms among older people living with HIV differently for men compared to women?

Researchers will compare a 12-week, twice a week remotely delivered tai chi/qigong intervention to a health education class of the same duration to determine if it improves depressive symptoms among older people living with HIV.

Participants will:

Attend either a tai chi/qigong class twice a week for 12 weeks or a health education class of the same duration delivered via Zoom. Each class will be 45-60 minutes in length.

Participate in 3 separate interviewer-administered interviews: at the time of enrollment, 3 months after the last class, and 9 months after the last class.

Keep a tracking log of their home practice of tai chi/qigong (only participants in the intervention group).

Use a biosensor (an earlobe sensor or chest strap) to measure their heart variability.

Go to their local lab (e.g., Quest or Labcorp) for blood draw at the time of enrollment and at 9 month post intervention (this will only be a subset of participants).

DETAILED DESCRIPTION:
Half of those living with HIV in the United States are over 50 years of age. As people living with HIV (PWH) live longer with the disease, the tradeoff is that they live with multiple comorbidities. One of the more common comorbidities is depression. There is a need to find innovative and accessible nonpharmacological interventions that can help older people living with HIV/AIDS to manage depressive symptoms that may also affect their treatment outcomes. Tai chi/Qigong (TCQ) is a series of slow, low-impact meditative movements that integrate breath work, meditation, and stances; and may improve depressive symptoms. Investigators propose testing the efficacy of a remotely delivered standardized TCQ intervention that has shown to be acceptable and feasible with a population of older people living with HIV/AIDS. Thus, this study proposes three aims: (i) to determine whether a remotely delivered TCQ intervention is directly efficacious in improving depressive symptoms compared to a health education control group among older PWH (50 years of age or older); (ii) to determine whether a remotely delivered TCQ intervention indirectly improves depressive symptoms via biological, psychological, and behavioral mechanisms compared to a health education control group among older PWH and (iii) to determine whether the direct and indirect associations between a TCQ intervention and depressive symptoms is moderated by gender among older PWH. Participants (n=326) will be recruited using social media sites (e.g., WebMD, google, Facebook) throughout the United States. All assessments will be conducted via Zoom videoconferencing or phone. Participants will be randomized to 1 of 2 conditions: the TCQ intervention, or a health education control group condition. Both the TCQ and the health education control condition will be delivered via Zoom to participants in the form of live, synchronous classes. Investigators will assess the efficacy of TCQ by looking at instruments that measure depression; and potential mechanisms such as sleep, fatigue, emotional regulation, and heart variability at baseline, 3-month, and 9-month post-intervention. Blood will also be collected at baseline and at 9-month to collect viral load and an inflammatory marker (C-reactive protein). Data will be described using descriptive techniques.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. The ability to provide consent assessed by the GAIN Cognitive Impairment Scale
2. Provision of signed and dated informed consent form
3. Must be 50 - 75 years old.
4. Must have been diagnosed with HIV by a healthcare professional (status confirmed at baseline by an uploaded picture of a recent lab report or medication bottle with name),
5. Must have reliable internet access,
6. Must have a smart phone
7. No substantial experience (regular weekly practice for more than 3 months in the past 12 months) with mind-body interventions,
8. Willing to participate for the length of the 12-week intervention and follow up assessments (a total of 12 months).
9. Must report stable housing for the past 60 days and the next 60 days;
10. Must have mild to moderate depressive symptoms (a score more than 5 but less than 19 on the PHQ-9 scale)
11. Must speak and understand English

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Reports high risk for suicide based on the CCSR screening tool.
2. Has participated in a study on mental health in the last 12 months.
3. Currently exercising at least 150 minutes a week

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms | Depressive symptoms will be assessed at enrollment (or baseline), 3 months post intervention, and 9 months post intervention.
  The 10-item Center for Epidemiologic Studies Depression Scale (CES-D) Short form will be used to assess depressive symptoms. Responses refer to the past week and range from: Rarely or none of the time (less than 1 day) = 0 to Most or all of the time (5-7 days) = 3. Scores range from 0-30 with greater scores meaning more depressive symptoms.

SECONDARY OUTCOMES:
Depressive symptoms | The Depression subscale of the DASS-21 will be assessed at enrollment (Baseline), at 3 month and at 9 months after the last class.
  Depressive symptoms will also be assessed using the Depression subscale from the Depression, Anxiety, Stress Scale (DASS-21). Responses refer to the past week and range from: Never=0 to Almost always=3. Higher scores mean more depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gladys E Ibanez, Ph.D., Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be electronic and stored in an open repository. Data include behavioral, psychological, and biological data collected at three different time points: baseline, 3 month and 9 month post intervention. This also includes the heart rate variability and blood collection results.
Supporting Information: Study Protocol
Time Frame: Data collected at baseline will be made available within 6 months of all baseline data being collected. Data collected at 3 month and 9 month post intervention will be made available 6 months after all data at that time point is collected.